CLINICAL TRIAL: NCT02888483
Title: PEAKS: Validation of Mobile Technologies for Clinical Assessment, Monitoring and Intervention
Brief Title: PEAKS: Validation of Mobile Technologies
Acronym: PEAKS
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Cancer Institute (NCI) (NIH); EveryFit, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB201600822 - N; 5R01AG042525-05 (NIH); SBIR HHSN261201500014C (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Health Services for Persons With Disabilities; Disability Evaluation; Exercise; Fitness Trackers; Validation Studies
Keywords: physical activity; energy expenditure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of this project is to evaluate and validate the accuracy and usability of a deployed beta sensor-based system. This is a cross-sectional validation study of 100 apparently health community dwelling adults aged 60+ years. Participants will perform standardized lifestyle, exercise and sedentary type physical activities in a clinic laboratory and home setting.

DETAILED DESCRIPTION:
Wearable activity monitors have the potential to continuously and objectively measure physical activity. However, existing monitors do not address the unique challenges that face older adults, who comprise the largest segment of population who suffer from physical disabilities and dexterity issues that can make using such monitors exceedingly difficult. In fact, the majority of wearable devices on the market address the needs of three broad segments:

1. Consumers: these devices are designed and optimized for motivated, healthy younger individuals and require pairing with smartphones to transmit data, while restricting or, at best, limiting access to raw data and algorithms.
2. Researchers: research-focused devices tend to be validated across a wide range of studies, but are not optimized for wearability or longitudinal use.
3. Developers: Developer-focused devices typically provide high configurability, a high- definition screen, and a variety of sensors (e.g. accelerometer, gyroscope, air pressure, light, temperature, etc.) that are suited for research and development, but are not optimized for power-efficient use.

To overcome the barriers that existing monitors impose on measuring free-living physical activity data, EveryFit developed in-home activity monitoring technology that addresses the specific and unique needs of the older population (incorporated in product called QMedic).

The overall objective of this project is to evaluate and validate the accuracy and usability of a deployed beta sensor-based system. The technology utilizes novel power-efficient engineering to continuously measure physical activity (including intensity, type and duration) in both laboratory and free-living settings. To accomplish this objective we will enroll 100 adults 60+ years of age who will perform standardized lifestyle, exercise and sedentary type physical activity in the laboratory. A subset of participants will also be asked to wear the monitor in free-living settings.

The proposed work can have far-reaching impact given the growth in the older adult population, which suffers disproportionally from chronic disease and functional impairments. Validating technology that measures physical activity continuously and accurately at the home is a critical step in scaling the system, conducting affordable population- scale studies, and maximizing the societal impact of the innovation.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ years old
* Community dwelling adults without significant health issues that would impact safety of participation
* Willingness to undergo all testing procedures
* Weight stable for at least three months
* Able to understand and speak English

Exclusion Criteria:

* Failure to provide informed consent
* Use of walker (use of a cane is permitted)
* Lower extremity amputation
* Develops chest pain or severe shortness of breath during physical stress
* Post-stroke syndrome causing ambulatory deficits (other stroke survivors permitted)
* Needs assistance with basic activities of daily living: feeding, dressing, continence, bathing, toileting, and transferring from a bed to a chair or from a chair to walking
* Lives in a nursing home; persons living in assisted or independent housing are not excluded
* Heavy drinking as drinking 5 or more drinks on the same occasion on each of 5 or more days in the past 30 days.
* For women who are child-bearing age (up to 62 years of age): pregnancy or breast-feeding
* Participation in a structured weight loss program or fad diet in the last month
* Weight reduction surgery in the past year
* Known neuromuscular disorder that restricts activity (e.g. Rhabdomyolysis, Myasthenia Gravis, Ataxia, Apraxia, post-polio syndrome, mitochondrial myopathy, etc.)
* Diagnosed neuropathy that causes pain that restricts activity
* Symptomatic peripheral arterial disease that restricts activity
* Unable to communicate because of severe hearing loss or speech disorder
* Severe visual impairment, which would preclude completion of the assessments
* Progressive, degenerative neurologic disease (e.g., Parkinson's Disease, Multiple Sclerosis, ALS)
* Severe rheumatologic or orthopedic diseases that significantly restricts activity (e.g., awaiting joint replacement, active inflammatory disease)
* Terminal illness, as determined by a physician
* Severe pulmonary disease, requiring the use of supplemental oxygen or steroid therapy
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, recent history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Other significant comorbid disease discovered during medical screening that would elicit safety concerns, (e.g. renal failure on hemodialysis, psychiatric disorder, chronic fatigue syndrome, etc.)
* Pacemakers and implanted cardiac defibrillators

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling population
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Metabolic equivalent (MET) value | within one month
  MET value of physical activities defined as the oxygen uptake (VO2 = milliliter• min-1•kg-1) during a steady state rate expressed as a function 3.5 milliliter• min-1•kg-1.

SECONDARY OUTCOMES:
Tradeoff Accuracy in metabolic equivalent estimation and power consumption | within one month
  We will manipulate the state machine that samples data from the device with different duty cycles based on contextual changes as measured by the accelerometer or classified by models that use the accelerometer data to classify behavior or categories of behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Manini, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Institute on Aging Clinical and Translational Research Building, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: University of Florida Institute on Aging — http://aging.ufl.edu/